CLINICAL TRIAL: NCT00294697
Title: Genetics of Innate Immune Response After Burn Trauma
Brief Title: Genetic Variation and Immune Responses After Injury
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Perry Adams, UT Southwestern Medical Center
Other Study IDs: 5K08GM071646-03 (NIH)
Record Dates: First submitted 2006-02-21; First posted 2006-02-22 (Estimated); Last update posted 2010-08-24 (Estimated); Status verified 2010-08

CONDITIONS: Sepsis; Pneumonia; Trauma; Burn; Injury
Keywords: polymorphisms; innate immune response; immunomonitoring; immuno paralysis
MeSH Terms: conditions — Sepsis; Pneumonia; Wounds and Injuries; Burns

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, Tissue, Fluids
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Our overall hypothesis is that genetic variations in innate immunity genes predispose patients to varying responses after injury by altering the systemic and local inflammatory responses. In addition, we hypothesize that these genetic differences are associated with different clinical outcomes

DETAILED DESCRIPTION:
The goal of this research proposal is to identify relationships that exist between specific genetic markers, immune responses to injury and infection (sepsis), and post injury clinical outcomes. Specifically, we will investigate the clinical impact of mutations involved in the innate immune response, which likely influence host response. To accomplish this goal we will collect and analyze data from patients with acute thermal injury, the most quantitative inflammatory stimulus experienced by humans. In addition, we propose to further characterize the immunologic response parameters to injury and infection, and their role in complicated sepsis. In this way, we will identify parameters associated with unfavorable clinical outcomes, and determine how these parameters differ among individuals with different genotypes. We propose to 1) evaluate associations between candidate SNPs within the NOD2/RIP2 signaling pathway and clinical outcome following burn injury, 2) evaluate the functional effects of alternate alleles at candidate SNPs; finally 3), we will use genetically engineered animal models to determine whether mutations in the NOD2 or RIP2 genes alter myocardial signal transduction mechanisms shown to play a role in myocardial inflammation/dysfunction after burn trauma. These approaches should allow us to evaluate more extensively clinically relevant interactions between specific genetic polymorphisms, the cellular expression of immune mediators, and burn-induced immune dysfunction. The proposed research should uncover genetic and/or acute immune-inflammatory parameters that identify patients who are at "high risk" and could as a result make possible the targeted design of pharmacologic intervention strategies that will inhibit the toxic effects of LPS and other bacterial pathogen components without paralyzing the host immunity of patients

ELIGIBILITY:
Inclusion Criteria: All burn,trauma, or acute surgery victims admitted to the surgical, burn or trauma units within 24 hours of injury will be considered for inclusion.

Exclusion Criteria:severe immunosuppression, DNR, severe trauma, terminal diseases.

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Burn, Trauma, and Surgical Patients
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2003-08; Study Completion 2011-10 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Fernando A Rivera-chavez, MD, Principal Investigator — Univ of Texas Southwestern Medical Center at Dallas
Locations (1):
- UT Southwestern Medical Center at Dallas, Dallas, Texas, United States

REFERENCES:
- [Background] Rivera-Chavez FA, Peters-Hybki DL, Barber RC, Lindberg GM, Jialal I, Munford RS, O'Keefe GE. Innate immunity genes influence the severity of acute appendicitis. Ann Surg. 2004 Aug;240(2):269-77. doi: 10.1097/01.sla.0000133184.10676.26. PMID 15273551
- [Background] Barber RC, Aragaki CC, Rivera-Chavez FA, Purdue GF, Hunt JL, Horton JW. TLR4 and TNF-alpha polymorphisms are associated with an increased risk for severe sepsis following burn injury. J Med Genet. 2004 Nov;41(11):808-13. doi: 10.1136/jmg.2004.021600. PMID 15520404
- [Background] Rivera-Chavez FA, Peters-Hybki DL, Barber RC, O'Keefe GE. Interleukin-6 promoter haplotypes and interleukin-6 cytokine responses. Shock. 2003 Sep;20(3):218-23. doi: 10.1097/01.shk.0000079425.52617.db. PMID 12923492
- [Background] Rivera-Chavez FA, Wheeler H, Lindberg G, Munford RS, O'Keefe GE. Regional and systemic cytokine responses to acute inflammation of the vermiform appendix. Ann Surg. 2003 Mar;237(3):408-16. doi: 10.1097/01.SLA.0000055274.56407.71. PMID 12616126